CLINICAL TRIAL: NCT00586885
Title: A Pilot Study: Therapeutic Effect of L-Alanine in Patients With Nonalcoholic Steatohepatitis
Brief Title: Effects of Alanine in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keith D Lindor, M.D. (Other)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Sponsor-Investigator, Keith D Lindor, M.D., Medical Doctor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1753-03
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; NASH; L-Alanine
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Alanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single arm, active treatment
  Interventions: Drug: L-alanine

INTERVENTIONS:
Drug: L-alanine — 6g of L-alanine (powder)once per day for the first month, twice per day for the second month, then three times per day from the third month for 10 months.

SUMMARY:
Purpose of this study is to assess the therapeutic efficacy of L-alanine in improving biological and histological findings by administrating 6-18g/day L-alanine for one year. We will also assess the safety and toxicity profile of long-term administration of L-alanine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age between 18 and 75
* Histological diagnosis of steatohepatitis with or without fibrosis made within one year of entry
* Transaminase levels (ALT or AST) more than 1.5 times the upper normal limit on at least two occasions with one assessment in three months or more prior to treatment of this study
* Previous and current alcohol consumption less than 20g per day by patient-provided information.
* Written informed consent specific for this protocol available prior to entry.
* Patients with diabetes and on stable medical management for six months prior to entry and an anticipated stable program throughout the study will be eligible. Medications that may be used include insulin, biguanides and sulfonylureas.
* Patients with congestive heart failure, hypertension and arrhythmia controlled by medications and without cardiac episodes during the past 6 months will be eligible.

Exclusion Criteria:

* Any causes for liver disease other than nonalcoholic steatohepatitis that are confirmed by patient history, laboratory data, or histological data
* Decompensated liver disease based on laboratory data, or clinical manifestations

  1. Hemoglobin <11.0g/dl for male, <10.0 g/dl for female
  2. White blood cells <2000 /mm3
  3. Platelet count <50,000/mm3
  4. Prothrombin time >INR 1.5
  5. Total Bilirubin >2.0 g/dl
  6. Albumin <3.0/dl
  7. The presence of ascites
  8. The presence of bleeding varices
  9. The presence of spontaneous encephalopathy
* Any previous experimental treatment of NASH within the past 3 months such as betaine, thiazolidinediones, α-tocopherol, or UDCA
* Pre-existing diseases/situations that could interfere with the results or the completion of this trial.
* Uncontrolled diabetes mellitus meeting following criteria in previous 3 months

  1. Fasting blood sugar >200 mg/dl
  2. Hemoglobin A1c >12%
* Renal or liver transplant patients
* Renal dysfunction in previous 3 months

  a) CCr <50ml/min
* Severe cardiovascular dysfunction in previous 6 months
* Congestive heart failure
* Uncontrolled hypertension
* Uncontrolled arrhythmia
* Patients with hyperlipidemia on a medical program for control of lipids which has had a change in drug treatment in the proceeding six months or with anticipated changes in the year of the study.
* Chronic pulmonary disease such as COPD requiring corticosteroid therapy in previous 3 months
* Active autoimmune or immunologically mediated diseases including systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel diseases in previous 12 months
* Previous (in three years) or present malignant disease except for non-melanoma skin cancer
* Untreated hyperthyroidism and hypothyroidism
* Substance abuse of oral, I.V., or inhaled drugs.
* If patients with history of substance abuse are considered as participants in this trial, patients must have abstained from using the abused substance for at least one year.
* Patients receiving methadone within the past 6 months are also excluded.
* Any other conditions that would make the patients unsuitable for enrollment in the opinion of the investigator in terms of interference in completing the trial and/or results of trial.
* Pregnant women
* Unwillingness of patients and /or partner to use contraceptive during treatment and for 3 months after discontinuation of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of long-term L-alanine supplementation and the therapeutic efficacy of long-term L-alanine supplementation by evaluating liver biochemistry and histological findings. | 1 year

SECONDARY OUTCOMES:
Determine the effect of L-alanine on gene profiles, anti-oxidant response and inflammatory response in hepatocytes. Evaluate possible correlation between therapeutic efficacy and gene profiles altered by L-alanine supplementation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Suzuki A, Charlton MR, Lymp JF, et al. A pilot study: No therapeutic effect of L-alanine in patients with nonalcoholic steatohepatitis. Food and Nutrition Sciences 2: 67-73, 2010.